CLINICAL TRIAL: NCT05203016
Title: Complications Associated With Intraoperative Hypothermia in Obstetrics and Plastic and Maxillofacial Surgery. Unicentric Cohort Study.
Brief Title: Complications Associated With Intraoperative Hypothermia.
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Other Study IDs: PI-3697
Record Dates: First submitted 2019-11-29; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2019-05

CONDITIONS: Hypothermia; Hemorrhage, Postpartum; Infection Surgical Wound; Transfusion-dependent Anemia
MeSH Terms: conditions — Hypothermia; Postpartum Hemorrhage; Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- caesarean sections
  Interventions: Other: Hipotermia/Normotermia
- Plastic surgery
  Interventions: Other: Hipotermia/Normotermia
- Maxillofacial surgery
  Interventions: Other: Hipotermia/Normotermia

INTERVENTIONS:
Other: Hipotermia/Normotermia — The temperature will be measured at the beginning and at the end of the surgery, as well as during admission to the Post-Anesthesia Care Unit, where the temperature normalization time will be noted in the event of hypothermia. In retrospect, those variables corresponding to the late postoperative period will be evaluated and the telephone interview will be conducted to assess the quality of care received. All the data will be reflected in the collection booklet that we present in the annex.

SUMMARY:
Maintaining intraoperative normothermia and temperature measurement is a marker of quality of care. We know that intraoperative hypothermia is associated with an increased risk of cardiovascular events, infection of the surgical wound, a longer hospital stay, discomfort, hemorrhage and transfusion demand.

Goals:

To know the incidence of perioperative hypothermia in routine clinical practice in different surgical settings in a national reference university hospital.

To establish if hypothermia is a risk factor for developing postoperative complications, focusing mainly on bleeding and infection of the surgical wound, in subjects aged between 18-65 years who come to the La Paz University Hospital for a surgical intervention in the Obstetrics / Plastic and Maxillofacial Surgery Services.

Hospital-based cohort study. A two-year follow-up of patients between 18 and 65 years will be carried out. Those patients with haemostasis disorders and infections in the preoperative period will be excluded.

Using a questionnaire on sociodemographic variables, the baseline conditions of the patients will be evaluated for inclusion in the study. Subsequently, the temperature will be measured at the beginning and at the end of the surgery, as well as during admission to the Post Anesthesia Care Unit, where the temperature normalization time will be noted in the event of hypothermia. In retrospect, those variables corresponding to the late postoperative period will be evaluated and the telephone interview will be conducted to assess the quality of care received. All the data will be reflected in the collection booklet that we present in the annex.

Patient demographics, case characteristics, and temperature records were summarized using descriptive statistics.

Microsoft Excel (Professional Plus 2010, version 14); it was used for data management and processing, with Stata (version 14; StataCorp LP, College Station, TX) for graphical representations and statistical tests. A multivariate analysis of potential confounding factors will be performed.

These results will serve to know the incidence of hypothermia according to the usual practice in a Spanish tertiary hospital and to establish recommendations in the management of intraoperative hypothermia and its prevention.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years, of any ethnic origin, with any type of comorbidities, with surgical indication in the Plastic, Maxillofacial and Obstetrics Surgery services scheduled or emergency under any mode of anesthesia (spinal, epidural, spinal combined or general anesthesia), following the usual practice of the service.
* That you agree to participate in the study by signing the informed consent.

Exclusion Criteria:

* Children under 18 or over 65 years of age, having received active prewarming in the preoperative period, received anti-fibrinolytic treatment, with bleeding diathesis, untreated perioperative anemia, preoperative perinatal infections and / or requiring intraoperative blood transfusion.
* Patients who for any reason should not be included in the study according to the evaluation of the research team and / or who refuse to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between 18 and 65 years old undergoing different types of surgeries (caesarean section / plastic and reparative / maxillofacial surgery) belonging to the Hospital Universitario la Paz will be monitored.
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Hypothermia | Through study completion, an average of 1 year.
  Body core temperature below 36ºC

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided